CLINICAL TRIAL: NCT04906993
Title: A Randomized, Open-Label, Controlled, Multi-Center Phase III Clinical Study of Camrelizumab Combined With Famitinib Malate Versus Platinum-based Chemotherapy in the Treatment of Recurrent/Metastatic Cervical Cancer
Brief Title: Camrelizumab Combined With Famitinib Malate for Treatment of Recurrent/Metastatic Cervical Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-329
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Platinum Compounds

STUDY DESIGN:
Intervention Model Description: 1:1 camrelizumab combined with famitinib malate platinum-based chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- camrelizumab combined with famitinib malate (Experimental)
  Interventions: Drug: camrelizumab； famitinib malate
- platinum-based chemotherapy (Active Comparator)
  Interventions: Drug: platinum-based chemotherapy

INTERVENTIONS:
Drug: camrelizumab； famitinib malate — Camrelizumab intravenously ; Famitinib Orally
  Arms: camrelizumab combined with famitinib malate
Drug: platinum-based chemotherapy — Physician's choice chemotherapy
  Arms: platinum-based chemotherapy

SUMMARY:
This study is a randomized, open-label, controlled, multi-center Phase III clinical study, aimed to evaluate the efficacy and safety of camrelizumab combined with famitinib malate versus platinum-based chemotherapy in the treatment of recurrent/metastatic cervical cancer. All enrolled patients will be randomly divided into 2 groups and continuously treated until any event that meets the criteria for end of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18-75 years (including 18 and 75 years, calculated based on the signing date of the informed consent)
2. Histopathologically confirmed recurrent/metastatic cervical squamous cell carcinoma that cannot be radically treated by surgery, radiotherapy or chemoradiotherapy
3. No prior systemic anti-cancer therapy for recurrent/metastatic disease
4. According to RECIST v1.1 criteria, the patient must have at least one measurable lesion
5. Able to normally swallow drug tablets
6. The organ function level is good
7. Willing to participate and able to comply with research programme requirements

Exclusion Criteria:

1. Has any malignancy <5 years prior to study entry.
2. Known to have brain or meningeal metastasis
3. Known to have autoimmune disease
4. Received live vaccinations 4 weeks before randomization or during the study period

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by the BIRC based on RECIST V1.1 criteria | up to 2 years
Overall survival (OS) | up to 3 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed by the investigator based on RECIST V1.1 criteria | up to 2 years
Objective response rate (ORR) assessed based on RECIST V1.1 criteria | up to 2 years
Disease control rate (DCR) assessed based on RECIST V1.1 criteria | up to 2 years
Duration of response (DOR) assessed based on RECIST V1.1 criteria | up to 2 years
Time to response (TTR) assessed based on RECIST V1.1 criteria | up to 2 years
Time to treatment failure (TTF) | up to 2 years
Progression-free survival (PFS) in subjects in the control group who receive camrelizumab after progression | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China